CLINICAL TRIAL: NCT07233863
Title: Effectiveness of Lymphovenous Bypass Procedure for Secondary Prevention of Lymphedema in Breast Cancer
Brief Title: Lymphovenous Bypass Procedure for Secondary Prevention of Lymphedema in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Principal Investigator, Bayu Brahma, MD, PhD, Dharmais National Cancer Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DP.04.03/11.5/095/2024
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema Arm
Keywords: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, pragmatic, parallel arm randomized clinical trial
Who Masked: Participant
Masking Description: Blinding is implemented in two conditions: the principal researcher (Bayu Brahma) will not know the patient's identity or medical history when assessing indocyanine green (ICG) lymphography results, and the patients will not see the type of treatment they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphovenous bypass (LVB) (Experimental): Sixty-eight subjects will be needed per group. LVB was performed by creating an intima-to-intima anastomosis between the afferent lymphatic vessels and the recipient veins. After surgery, follow-up will be done every 6 months for 2 years. During follow-up, a comprehensive evaluation will be performed, including history and physical examinations, radiological and histopathological examinations, UEL index, ICG lymphography, and quality-of-life evaluation. Each subject will complete the Lymphedema Quality of Life Questionnaire.
  Interventions: Procedure: Lymphovenous bypass (LVB)
- Physiotherapy (No Intervention): Sixty-eight subjects will be needed per group. Patients will receive physiotherapy from trained physiotherapists. The protocol includes manual lymphatic drainage (massage techniques), compression, skin care, and arm exercises. Follow-up will be done every 6 months for 2 years. During follow-up, a comprehensive evaluation will be performed, including history and physical examinations, radiological and histopathological examinations, UEL index, ICG lymphography, and quality-of-life evaluation. Each subject will complete the Lymphedema Quality of Life Questionnaire.

INTERVENTIONS:
Procedure: Lymphovenous bypass (LVB) — The Lymphovenous Bypass (LVB) procedure in this study is a microsurgical supermicrosurgery-based intervention specifically designed for the secondary prevention of breast cancer-related lymphedema following axillary lymph node dissection.
  Arms: Lymphovenous bypass (LVB)

SUMMARY:
This study aims to evaluate the effectiveness of the Lymphovenous Bypass (LVB) procedure compared to physiotherapy alone as secondary prevention of lymphedema in breast cancer patients undergoing axillary lymph node dissection.

DETAILED DESCRIPTION:
In the intervention group, LVB was performed with intima-to-intima coaptation using the super microsurgery technique. The anastomosis was between the afferent lymphatic vessel and the recipient vein. The upper extremity lymphedema (UEL) index and indocyanine green (ICG) lymphography are utilized to evaluate the progression of lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients aged ≥ 18 years with an ECOG score > 1
* Breast cancer patients with post-axillary lymph node dissection diagnosed with stage 0 and I lymphedema.
* Those who have never undergone lymphedema physiotherapy.

Exclusion Criteria:

* Patients with dermal backflow before axillary lymph node dissection (ALND).
* Patients with breast cancer lymphedema who are unable to undergo a 24-month follow-up at Dharmais Cancer Hospital.
* Patients with iodine allergy, severe asthma, decreased kidney function, pregnancy, or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2027-03-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
BCRL improvement rate | 24 months
  BCRL definition:
  Post-operation subject condition with the presence of minimum DB 2 with one or both symptoms (swelling, heaviness), and an increment of UEL index >10% compared to pre-operation OR Post-operation subject condition with presence of ≥ DB 2 with minimum area 30% in one arm region in one of the arm lymphatic pathways (anterior or posterior), without presence of symptoms (swelling or heaviness), and increment of UEL index >10% compared to pre-operation.
  International Society of Lymphology (ISL) stage 1 definition:
  An early stage of lymphedema is characterized by soft tissue swelling that may subside with limb elevation or overnight rest, without permanent structural changes.
  BCRL improvement :
  Improvement in ICG lymphography stage with or without clinical signs (UEL <10% and or symptoms improvement)

SECONDARY OUTCOMES:
Quality of life in lymphedema | 24 months
  QLQ-BR23 is a supplement to the EORTC QLQ-30, specific to breast cancer patients, containing 23 questions and scored from 0 (not at all) to 4 (very much). To evaluate the quality of life, we asked three questions about the arm (pain, swelling, and mobility issues). The quality of life decreases with a higher score.
Adverse event of lymphedema | 24 months
  Complications such as seroma, hematoma, wound separation, bleeding, and wound infection can be seen after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bayu Brahma, MD, PhD, Principal Investigator — Dharmais Cancer Hospital - National Cancer Center
Locations (1):
- Dharmais National Cancer Center, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koshima I, Inagawa K, Urushibara K, Moriguchi T. Supermicrosurgical lymphaticovenular anastomosis for the treatment of lymphedema in the upper extremities. J Reconstr Microsurg. 2000 Aug;16(6):437-42. doi: 10.1055/s-2006-947150. PMID 10993089
- [Result] Brahma B, Putri RI, Reuwpassa JO, Tuti Y, Alifian MF, Sofyan RF, Iskandar I, Yamamoto T. Lymphaticovenular Anastomosis in Breast Cancer Treatment-Related Lymphedema: A Short-Term Clinicopathological Analysis from Indonesia. J Reconstr Microsurg. 2021 Oct;37(8):643-654. doi: 10.1055/s-0041-1723940. Epub 2021 Mar 1. PMID 33648010
- [Result] Agarwal S, Garza RM, Chang DW. Lymphatic Microsurgical Preventive Healing Approach (LYMPHA) for the prevention of secondary lymphedema. Breast J. 2020 Apr;26(4):721-724. doi: 10.1111/tbj.13667. Epub 2019 Oct 20. PMID 31631442